CLINICAL TRIAL: NCT06072677
Title: Probing the Neurophysiological Mechanisms Underlying Sex-specific Testosterone-mood Relationships During Puberty: A Randomized Controlled Trial Using a Smartphone-based Training Program
Brief Title: Adolescent Mood During Puberty and Testosterone
Acronym: AMPT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Foundation of Hope, North Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 23-1336
Record Dates: First submitted 2023-10-02; First posted 2023-10-10 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Adolescent Depression
Keywords: Puberty; Depression; Mood disturbance; Adolescence; Stress; Peripubertal Transition; Hormones; EEG; Sex differences
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Minds Program (Experimental): Participants in this group will begin the Healthy Minds Program immediately following the 4-week baseline period.
  Interventions: Behavioral: Healthy Minds Program
- Waitlist Control (Other): After the 4-week baseline period, participants in the waitlist control condition will wait an additional 4 weeks before starting the Healthy Minds Program.
  Interventions: Behavioral: Healthy Minds Program

INTERVENTIONS:
Behavioral: Healthy Minds Program — The Healthy Minds Program is a 4-week mobile program to improve coping and emotion regulation skills. It includes 4 training modules corresponding to key pillars of wellbeing: awareness(focused attention/awareness of thoughts/emotions), connection (empathy, compassion, social connection), insight (clarity of identify/experience) and purpose (applying values/motivations). The Healthy Minds Program includes 2 introductory audio lessons and guided meditations, and each 1-week module includes 2 podcast lessons (5-7 minutes) with psychoeducation and practical examples, and 3 guided meditations relevant to the module topic, for a total of 10 lessons and 14 guided meditations.

SUMMARY:
Starting at puberty, female adolescents are nearly three-times more likely to develop internalizing disorders, like depression, while male adolescents are two-times more likely to develop externalizing disorders, like attention deficit hyperactivity disorder (ADHD). This divergence between the sexes during puberty suggests sex-specific pathways of risk and differential effects of sex hormones. The purpose of this research is to determine: 1) sex-specific neural and endocrine features of the pubertal transition that may mediate sex differences in adolescent mood disorders, and 2) the neurophysiological basis of susceptibility to hormone change during puberty.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 11 and 14
* Have their own personal mobile device and capability to download the MyCap and Healthy Minds apps
* Experienced a stressful life event within the last year, or endorse moderate depression (defined by a CES-DC score 16 or higher)

Exclusion Criteria:

* Previous experience with the Healthy Minds Program
* Regular meditation practice
* Current or history of manic episodes, psychotic symptoms, or current suicidal intent
* Taking any form of exogenous hormones or intrauterine device (IUD) within one month of participation in the study
* Taking medications that directly alter cardiovascular or neurological function

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-08-24 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
CES-DC Score Over Time | up to Week 8
  The 20-item Center for Epidemiological Studies Depression Scale for Children (CES-DC) will be the primary measure of severity of depressive symptoms. Each item is rated 0 (not at all) to 3 (a lot), with items 4, 8, 12, and 16 being reversed scored. The total CES-DC score may range from 0-60. Higher scores indicate more severe depressive symptoms. Scores of 15 or greater are suggestive of significant depressive symptoms. The overall CES-DC score will be assessed at the end of each week in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Andersen, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Carolina Crossing B, Suite 1, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP
Time Frame: beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.